CLINICAL TRIAL: NCT05797714
Title: A Prospective, Randomized, Blank Control, Multicenter Study to Evaluate the Efficacy and Safety of Alanine Aminotransferase（TMF）in the Treatment of Chronic Hepatitis B Patients With Normal Alanine Aminotransferase.
Brief Title: The Effectiveness and Safety of TMF in the Treatment of Chronic Hepatitis B Patients With Normal ALT.
Acronym: Promote
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Promote
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: HBV Infection; Chronic Hepatitis b
Keywords: Normal Alanine Aminotransferase; Treatment; Effectiveness; Safety
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Intervention Model Description: The subjects were randomly divided into two groups. One group received TMF treatment for 48 weeks. Aonther group received no antiviral therapy and served as a blank control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMF treatment group (Experimental): TMF 25mg QD, from baseline to 240 weeks
  Interventions: Drug: Tenofovir Amibufenamide（TMF）
- Blank control group (No Intervention): No antiviral therapy is given. If ALT>2 ULN (40 IU/L) for HBeAg-positive patients or > ULN for HBeAg-negative patients during the study period, blank control group can be switched to TMF treatment once a day, 25mg/ time orally until the end of the study.

INTERVENTIONS:
Drug: Tenofovir Amibufenamide（TMF） — TMF, 25mg QD, from baseline to 240 weeks
  Other Names: HengMu
  Arms: TMF treatment group

SUMMARY:
This is a multicenter, randomized, open, blank controlled trial ，in order to evaluate the effectiveness and safety of Amibufenamide（TMF） in the treatment of chronic hepatitis B virus infection patients with normal ALT .

DETAILED DESCRIPTION:
Although the indications for antiviral therapy for patients with chronic hepatitis B have been gradually expanded in different guidelines, antiviral treatment efficacy remains unclear among patients with alanine aminotransferase (ALT) < 1 upper limits of normal (ULN). This study aimed to evaluate the the effectiveness and safety of TMF for these patients.

Tenofovir amibufenamide (TMF; codename: HS-10234), another formulation of tenofovir, shared the same ProTide technology as tenofovir alafenamide, which can provide more efficient intracellular delivery than TDF.

ELIGIBILITY:
Inclusion Criteria:

1. Must have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study screening.
2. Male and non-pregnant, non-lactating females, from 18 up to 65 years of age (based on the date of the screening visit). A negative serum pregnancy test at screening is required for female subjects of childbearing potential.
3. Documented evidence of chronic HBV infection (e.g. HBsAg positive for more than 6 months).
4. Normal alanine aminotransferase: serum HBV DNA >20 IU/mL and serum ALT level ≤ULN (40 IU/L) during screening.
5. Treatment-naive subjects will be eligible for enrollment.
6. Must be willing and able to comply with all study requirements.

Exclusion Criteria:

1. Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study.
2. Males and females of reproductive potential who are unwilling to use an "effective", protocol specified method(s) of contraception during the study.
3. Co-infection with HCV virus, HIV, HEV or HDV or combined with autoimmune liver disease, metabolism-related fatty liver disease, drug-induced liver injury;
4. Evidence of hepatocellular carcinoma (e.g. as evidenced by recent imaging).
5. Any history of, or current evidence of, clinical hepatic decompensation (e.g. ascites encephalopathy or variceal hemorrhage) or liver stiffness over 9kpa measured by TE.
6. Abnormal hematological and biochemical parameters, including:

   Hemoglobin < 10 g/dl Absolute neutrophil count < 0.75 × 10^9/L Platelets ≤ 50 × 10^9/L AST > 10 × ULN Total Bilirubin > 2.5 × ULN Albumin < 3.0 g/dL INR > 1.5 × ULN (unless stable on anticoagulant regimen) eGFR<50mL/min
7. Received solid organ or bone marrow transplant.
8. Malignancy within the 5 years prior to screening, with the exception of specific cancers that are cured by surgical resection (basal cell skin cancer, etc).
9. Currently receiving therapy with immunomodulators (e.g. corticosteroids), investigational agents, nephrotoxic agents, or agents capable of modifying renal excretion.
10. Complicated with uncontrollable cardiovascular and cerebrovascular diseases.
11. Subjects on prohibited concomitant medications. Subjects on prohibited medications, otherwise eligible, will need a wash out period of at least 30 days,Known hypersensitivity to study drugs, metabolites, or formulation excipients.
12. Current alcohol or substance abuse judged by the investigator to potentially interfere with participant compliance.
13. Any other clinical condition or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with dosing requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation the percentage of Participants with Hepatitis B Virus (HBV) DNA < 20 IU/mL | Week 48
  The primary efficacy endpoint was the proportion of patients with HBV DNA < 20 IU/mL at week 48

SECONDARY OUTCOMES:
Evaluation the change from Baseline in HBV DNA | Week 48，Week 96，Week 144，week 240
  Change from baseline in HBV DNA
Evaluation the proportion of Patients Achieving Hepatitis B Surface Antigen (HBsAg) Loss | Week 48，Week 96，Week 144，Week 240
  Proportion of patients achieving Hepatitis B surface antigen (HBsAg) loss
Evaluation the proportion of Patients Achieving HBsAg Seroconversion | Week 48，Week 96, Week 144, Week 240
  Proportion of patients achieving HBsAg seroconversion
Evaluation the proportion of Patients Achieving HBeAg Seroconversion | Week 48，Week 96，Week 144, Week 240
  Proportion of patients achieving HBeAg seroconversion
Evaluation the proportion of Patients Achieving HBeAg Loss | Week 48，Week 96，Week 144 ，Week 240
  Proportion of patients Achieving HBeAg Loss
Evaluation the change from Baseline in HBsAg | Week 48，Week 96，Week 144，Week 240
  Change from baseline in HBsAg
Evaluation the percentage of Participants with resistance | Week 48，Week 96，Week 144，Week 240
  Percentage of participants with resistance
Evaluation the change from Baseline in liver fibrosis | Week 48，Week 96，Week 144，Week 240
  Change from baseline in liver fibrosis
Evaluation the proportion of Patients with get hepatitis acute attack（ALT >5 ULN (40 IU/L)） | Week 48，Week 96，Week 144，Week 240
  Proportion of patients with get hepatitis acute attack（ALT >5 ULN (40 IU/L)）
Evaluation the percentage of Participants with Hepatitis B Virus (HBV) DNA < 20 IU/mL | Week 96，Week 144，Week 240
Evaluation the change from Baseline in Bone biomarker（β-CTX and P1NP） | Week 48，Week 96，Week 144，Week 240
Evaluation the change from Baseline in sCR | Week 48，Week 96，Week 144，Week 240
AE ,SAE | Week 48，Week 96，Week 144，Week 240
The proportion of subjects with liver-related events | Week 48，96，144，192，240
  Liver decompensation, acute-on-chronic liver failure, hepatocellular carcinoma, liver transplantation, all-cause mortality

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - The Second Xiangya Hospital, Central South University, Changsha, Hunan
  - Beijing You'An Hospital, Capital Medical University, Beijing
  - People's Hospital of Dongyang City, Dongyang
  - Fuyang Second People's Hospital, Fuyang
  - The First People's Hospital of Xiaoshan District, Hangzhou, Zhejiang Province, Hangzhou
  - LiShui People's Hospital of Zhejiang Province, Lishui
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjin
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China., Shanghai
  - Shanghai East Hospital, Shanghai
  - The Fifth People's Hospital of Suzhou, Suzhou
  - The Fifth People's Hospital of Wuxi, Wuxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu Z, Jin Q, Zhang Y, Gong G, Wu G, Yao L, Wen X, Gao Z, Huang Y, Yang D, Chen E, Mao Q, Lin S, Shang J, Gong H, Zhong L, Yin H, Wang F, Hu P, Xiao L, Li C, Wu Q, Sun C, Niu J, Hou J; TMF Study Group. Randomised clinical trial: 48 weeks of treatment with tenofovir amibufenamide versus tenofovir disoproxil fumarate for patients with chronic hepatitis B. Aliment Pharmacol Ther. 2021 Nov;54(9):1134-1149. doi: 10.1111/apt.16611. Epub 2021 Sep 29. PMID 34587302
- [Result] Gui H, Shen Y, Tan L, Hu P, Qian F, Wu X, Qiu Y, Zheng S, Lv J, Shi Y, Li J, Jiang Y, Hu Z, Nie F, Huo Y, Qu L, Xie Q. Interim Analysis of 48-week Tenofovir Amibufenamide Treatment in Chronic Hepatitis B Patients with Normal Alanine Aminotransferase Levels: The PROMOTE Study. J Clin Transl Hepatol. 2025 Jul 28;13(7):568-577. doi: 10.14218/JCTH.2025.00162. Epub 2025 Jun 30. PMID 40937079
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40937079/